CLINICAL TRIAL: NCT06428461
Title: Evaluation of Supraclavicular Brachial Plexus Blocks At Different Volumes Under Ultrasound Guidance in Upper Extremity Surgery and Their Impact on Optic Nerve Sheath Diameter
Brief Title: Evaluation of Supraclavicular Brachial Plexus Blocks At Various Volumes: Impact on Optic Nerve Sheath Diameter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, ismet çopur, Investigator - Medical doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: PAU-ANEST-RHE-IC-01
Record Dates: First submitted 2024-05-14; First posted 2024-05-24 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Upper Limb Injury; Intracranial Pressure Increase
Keywords: Supraclavicular brachial plexus block; Intracranial pressure; Optic nerve sheath diameter
MeSH Terms: conditions — Arm Injuries; Intracranial Hypertension | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: Four different volumes will be administered for the supraclavicular block:
  1. For the control group, we plan to use a mixture of 7.5 mL of 0.5% bupivacaine (BUVICAINE-POLIFARMA-TEKIRDAG) and 7.5 mL of 2% prilocaine (PRILOC-VEM İlaç San. ve Tic. A.Ş. Kapaklı/TEKIRDAĞ) for a total of 15 mL.
  2. For the research group, we plan to use a mixture of 10 mL of 0.5% bupivacaine and 10 mL of 2% prilocaine for a total of 20 mL.
  3. For the research group, we plan to use a mixture of 12.5 mL of 0.5% bupivacaine and 12.5 mL of 2% prilocaine for a total of 25 mL.
  4. For the research group, we plan to use a mixture of 15 mL of 0.5% bupivacaine and 15 mL of 2% prilocaine for a total of 30 mL.
  Glob axis and optic nerve sheath diameter measurements for both eyes will be re-measured and recorded using B-mode ultrasound at 20 and 60 minutes after the supraclavicular block.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Total of 15 mL. (Active Comparator): For the control group, we plan to use a mixture of 7.5 mL of 0.5% bupivacaine (BUVİCAİNE®) and 7.5 mL of 2% prilocaine (PRİLOC®) for a total of 15 mL. single shot supraclavicular brachial plexus block.
  Interventions: Procedure: Supraclavicular brachial plexus block; Device: Measurement of Optic Nerve Sheath Diameter (ONSD) Using B-Mode Ultrasound; Device: Assessment of Peripheral Nerve Block Success Using Perfusion Index Measurement; Device: End-Tidal Carbon Dioxide (EtCO2) Measurement
- Total of 20 mL. (Active Comparator): For the research group, we plan to use a mixture of 10 mL of 0.5% bupivacaine (BUVİCAİNE®) and 10 mL of 2% prilocaine (PRİLOC®) for a total of 20 mL.
  Interventions: Procedure: Supraclavicular brachial plexus block; Device: Measurement of Optic Nerve Sheath Diameter (ONSD) Using B-Mode Ultrasound; Device: Assessment of Peripheral Nerve Block Success Using Perfusion Index Measurement; Device: End-Tidal Carbon Dioxide (EtCO2) Measurement
- Total of 25 mL. (Active Comparator): For the research group, we plan to use a mixture of 12.5 mL of 0.5% bupivacaine (BUVİCAİNE®) and 12.5 mL of 2% prilocaine (PRİLOC®) for a total of 25 mL.
  Interventions: Procedure: Supraclavicular brachial plexus block; Device: Measurement of Optic Nerve Sheath Diameter (ONSD) Using B-Mode Ultrasound; Device: Assessment of Peripheral Nerve Block Success Using Perfusion Index Measurement; Device: End-Tidal Carbon Dioxide (EtCO2) Measurement
- Total of 30 mL. (Active Comparator): For the research group, we plan to use a mixture of 15 mL of 0.5% bupivacaine (BUVİCAİNE®) and 15 mL of 2% prilocaine (PRİLOC®) for a total of 30 mL.
  Interventions: Procedure: Supraclavicular brachial plexus block; Device: Measurement of Optic Nerve Sheath Diameter (ONSD) Using B-Mode Ultrasound; Device: Assessment of Peripheral Nerve Block Success Using Perfusion Index Measurement; Device: End-Tidal Carbon Dioxide (EtCO2) Measurement

INTERVENTIONS:
Procedure: Supraclavicular brachial plexus block — A supraclavicular brachial plexus block will be performed under ultrasound guidance. The patient will be taken to the preoperative block room, positioned supine with the bed elevated at a 30° angle, and the head turned away from the arm being blocked. To avoid intraneural injection, the block will use both ultrasound and a nerve stimulator (Plexygon, Vygon-Italy) with a 22G 50 mm 20° stimulating needle (Echoplex, Braun-France). A low-frequency ultrasound probe will be placed above the clavicle to visualize the subclavian artery and vein. Using an in-plane approach, the needle will be inserted laterally to medially from the mid-clavicular point through the skin and subcutaneous tissue. Under ultrasound guidance, the needle will be advanced towards the anatomical corner where the brachial plexus and subclavian artery are adjacent (corner pocket), and a local anesthetic agent will be injected to perform the block.
Device: Measurement of Optic Nerve Sheath Diameter (ONSD) Using B-Mode Ultrasound — Before the block, both eyes will be measured for optic nerve sheath diameter (ONSD) using B-mode ultrasound (USG) with a GE LOGIQ E device. The patient will be supine with the bed elevated at a 30° angle, eyes closed, and a protective barrier applied. Both globes will be filled with water-soluble ultrasound gel, and imaging will be done with a 7.5 MHz linear probe at a 7 cm depth. For transverse ONSD measurement, the probe will be placed transversely in the coronal plane, with the marker notch pointing right. When the optic nerve entry into the globe is clear, transverse ONSD will be measured 3 mm below. For sagittal measurement, the probe will be placed sagittally in the coronal plane, with the marker notch pointing towards the body. Sagittal ONSD will be measured 3 mm below the entry point. Both internal and external diameters of the optic nerve sheath will be measured in transverse and sagittal planes, and the transverse diameter of the globe will also be measured.
Device: Assessment of Peripheral Nerve Block Success Using Perfusion Index Measurement — Investigator plan to measure the Perfusion Index (PI) as an objective method for determining the success of peripheral nerve blocks, different from traditional tests. PI is an indicator of peripheral perfusion that can be continuously measured non-invasively with a pulse oximeter. PI represents the ratio of pulsatile blood flow to non-pulsatile blood flow in peripheral tissue. The Mindray uMEC 12 device will be used for this measurement.
Device: End-Tidal Carbon Dioxide (EtCO2) Measurement — End-tidal carbon dioxide (EtCO2) measurement: The Medtronic Capnostream 35 device will be used for EtCO2 measurements. All patients will receive oxygen support at a rate of 1-2 L/min. If peripheral oxygen saturation falls below 95%, oxygen support will be increased to 3-6 L/min via nasal cannula.

SUMMARY:
This study aimed to evaluate the anesthesia adequacy, side effects, and complication rates, as well as the postoperative pain relief effectiveness of supraclavicular brachial plexus blocks administered at different volumes under ultrasound guidance. Additionally, the investigators utilized ultrasound to measure optic nerve sheath diameters and investigated their relationship with intracranial pressure across varying block volumes.

DETAILED DESCRIPTION:
Regional anesthesia involves temporarily blocking nerve transmission and pain sensation in specific areas of the body without causing loss of consciousness. Regional anesthesia techniques include peripheral nerve blocks (PNB), topical anesthesia, infiltration anesthesia, regional intravenous anesthesia (RIVA), and neuroaxial blocks (spinal and epidural anesthesia).

Brachial plexus blocks are among the most commonly used regional anesthesia methods within peripheral nerve block applications. Peripheral nerve blocks of the upper extremity can be used either alone for surgical anesthesia or added to general anesthesia for postoperative pain control. Brachial plexus blocks can be performed using various approaches including interscalene, supraclavicular, infraclavicular, and axillary approaches.

The supraclavicular block aims to effectively control pain through a procedure targeting the shoulder and upper extremity nerves known as the brachial plexus. Complications of supraclavicular blocks may include pneumothorax secondary to lung trauma, hoarseness due to ipsilateral recurrent laryngeal nerve blockade, Horner syndrome due to stellate ganglion blockade, and hemidiaphragmatic paralysis due to phrenic nerve blockade. The incidence and severity of these complications are reduced with the use of ultrasound (USG) guidance and low-volume techniques.

Intracranial pressure (ICP) refers to the pressure formed by the brain and spinal fluid, tissues, and blood surrounding the brain and spinal cord. Normally ranging between 5-15 mmHg, this pressure is critical for brain function and circulation. Abnormal increases in intracranial pressure can lead to intracranial hypertension, with main causes including brain tumors, edema, head trauma, brain aneurysms, intracranial hemorrhage, and issues related to the production and drainage of cerebrospinal fluid. External ventricular drainage (EVD) catheterization is the gold standard method for evaluating increased intracranial pressure. Measurement of optic nerve sheath diameter (ONSD) has been described as a valuable diagnostic method in clinical applications for evaluating intracranial pressure.

Observational studies have shown that in cervical sympathetic blocks and interscalene blocks, indirect increases in intracranial pressure can be demonstrated through ultrasound (USG) measurements of optic nerve sheath diameter. It has been shown that hemidiaphragmatic paralysis due to ipsilateral phrenic nerve involvement, which is frequently seen in interscalene brachial plexus blocks, also occurs in supraclavicular brachial plexus blocks in a volume-dependent manner. There are studies in the literature on supraclavicular block applications with different volumes and doses. However, the investigators have not come across a study evaluating the clinical outcomes of optic nerve sheath diameter measurement along with anesthesia quality, side effects, and complications in ultrasound-guided supraclavicular blocks at different volumes.

In this study, the investigators aimed to evaluate the anesthesia adequacy, side effects, and complication rates, as well as the postoperative analgesic efficacy of supraclavicular brachial plexus blocks performed at different volumes in our clinical practice under ultrasound guidance. Additionally, the investigators aimed to measure optic nerve sheath diameters with ultrasound and establish their relationship with intracranial pressure according to these different volumes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 50, of both genders, with planned surgery on the finger, wrist, elbow joint, and distal region, and classified as ASA I-II, will be included in the study. In this study, patients will be informed about the anesthesia method and the tests to be conducted, and those who consent will be asked to sign an informed consent form as voluntary participants.

Exclusion Criteria:

* Patients who do not accept the procedures and tests
* Those with diseases that may cause increased intracranial pressure
* Patients with severe heart failure
* Patients with second or third degree atrioventricular block
* Patients with unstable angina history
* Patients with COPD and chronic asthma
* Patients with a history of myocardial infarction (MI) within the last 6 weeks
* Patients with a heart rate below 50 beats/min
* Patients with systolic blood pressure below 90 mmHg
* Patients with liver failure
* Patients with kidney failure
* Patients for whom supraclavicular block anatomically cannot be performed
* Those with neurological or psychological diseases that make it difficult to assess the tests
* Patients allergic to any of the study drugs
* Pregnant women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-11-03 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter measured by ultrasonography | Before block, After block 20 minutes, After block 60 minutes
  Optic nerve sheath diameter will be measured using B-mode ultrasonography.

SECONDARY OUTCOMES:
Perfusion index (PI) | The PI values will be measured and recorded at 0, 2, 4, 6, 8, 10, 15, 20, and 25 minutes in both arms.
  PI, an objective method different from traditional tests, to determine the success of peripheral nerve block. PI is an indicator of peripheral perfusion that can be measured continuously and non-invasively with a pulse oximeter. PI is the ratio of pulsatile blood flow to non-pulsatile blood flow in peripheral tissue. Its normal value ranges from 0.02 to 20. After peripheral nerve block, vasodilation occurs in the vessels due to sympathetic blockade, resulting in an increase in PI values, which occurs earlier than motor and sensory block. PI monitoring provides more objective results for evaluating the onset of the block. The cut-off value indicating that the block is successful is a PI increase to 3.03 times the baseline value 10 minutes after the block is administered.
Non-invazive end-tidal carbon dioxide (EtCO2) | EtCO2 will be measured and recorded at 0, 10, 20, 30, 60 minutes, and at the end of surgery after the block is performed.
  Non-invasive EtCO2 measurement is a method used to monitor the concentration of carbon dioxide (CO2) at the end of expiration.
Pinprick test | The pinprick test will be evaluated 5 minutes after the block is performed and subsequently at 5-minute intervals, up to a maximum of 30 minutes. The results will be recorded throughout these evaluations.
  The pinprick test is a clinical procedure used to evaluate sensory nerve function. A small, sharp object, such as a pin or needle, is gently pressed against the skin to assess the patient's ability to feel pain.
Modified Bromage Scale | The Modified Bromage Scale will be evaluated 5 minutes after the block is performed and subsequently at 5-minute intervals, up to a maximum of 30 minutes. The results will be recorded throughout these evaluations.
  The Modified Bromage Scale is a clinical tool used to assess the degree of motor block in patients who have received regional anesthesia. The scale ranges from 0 to 3, with each level indicating a different degree of motor impairment:
  * 0: No motor block; full flexion of knees and feet.
  * 1: Partial motor block; able to move knees but not feet.
  * 2: Almost complete motor block; able to move feet only.
  * 3: Complete motor block; unable to move knees or feet.
Verbal Pain Score | The Verbal Pain Score will be assessed at the following intervals after surgery: immediately in the recovery room, at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, and 24 hours postoperatively.
  The Verbal Pain Score is a subjective measure used to assess a patient's level of pain. Patients are asked to rate their pain on a scale from 0 to 10, where 0 indicates no pain and 10 represents the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Rıza Hakan Erbay, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gundogdu O, Avci O. Evaluation of the Effect of Interscalene Brachial Plexus Block on Intracranial Pressure Using Optic Nerve Sheath Diameter and Internal Jugular vein Collapsibility Index. J Coll Physicians Surg Pak. 2022 Oct;32(10):1249-1254. doi: 10.29271/jcpsp.2022.10.1249. PMID 36205266
- [Background] Pansell J, Bell M, Rudberg P, Friman O, Cooray C. Optic nerve sheath diameter measurement by ultrasound: Evaluation of a standardized protocol. J Neuroimaging. 2022 Jan;32(1):104-110. doi: 10.1111/jon.12936. Epub 2021 Sep 23. PMID 34555223
- [Background] Hylkema C. Optic Nerve Sheath Diameter Ultrasound and the Diagnosis of Increased Intracranial Pressure. Crit Care Nurs Clin North Am. 2016 Mar;28(1):95-9. doi: 10.1016/j.cnc.2015.10.005. Epub 2015 Dec 23. PMID 26873762